CLINICAL TRIAL: NCT00699933
Title: Diagnostic and Interventional Therapy in Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Dr. Tanja Brünnler, University of Regensburg
Other Study IDs: 08/008
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2010-06

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; interventional therapy; CT-guided drainage therapy; percutaneous necrosectomy; Comparison of different diagnostic procedures: MRI, CT, Ultrasound; Evaluation of interventional therapy including percutaneous drainage techniques und necrosectomies
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Evaluation of one study cohort
  Interventions: Other: CT-guided percutaneous drainage technique

INTERVENTIONS:
Other: CT-guided percutaneous drainage technique — Evaluation of different diagnostics and evaluation of outcome of patients who received percutaneous CT-guided drainage for necrotic debridement and analyze the further outcome

SUMMARY:
The study aims to evaluate the course of patients with acute pancreatitis. Thereby we analyze different diagnostics and compare ultrasound, MRI and CT-scan in detection of necrotic areas and evaluate interventional therapy methods like percutaneous drainage techniques regarding the outcome. Laboratory values were assessed as well.

DETAILED DESCRIPTION:
For laboratory values different inflammation markers were measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Acute pancreatitis
* Written formal consent

Exclusion Criteria:

* Pregnancy
* Missing formal consent
* Individual contraindications for CT-scan
* MRI or endoscopic ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | weekly

SECONDARY OUTCOMES:
time to surgery | weekly
active necrosectomy | weekly
ICU stay | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Schölmerich, Prof., Study Director — Director of Department of Internal Medicine I; Stefan Feuerbach, Prof., Study Director — Director of Department of Radiology
Locations (1):
- Department of Internal medicine I, University of Regensburg, Regensburg, Germany